CLINICAL TRIAL: NCT00423813
Title: A Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study of Xyrem® (Sodium Oxybate) in Subjects With Fibromyalgia.
Brief Title: A Safety and Efficacy Study of Xyrem® (Sodium Oxybate) to Treat Fibromyalgia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-009
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2011-12

CONDITIONS: Fibromyalgia
Keywords: FMS; Fibro; pain; Body pain; tenderness; stiffness; muscular pain; joint pain
MeSH Terms: conditions — Fibromyalgia; Pain; Myalgia; Arthralgia | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: Xyrem®

INTERVENTIONS:
Drug: placebo — Oral Solution
  Arms: 1
Drug: Xyrem® — two doses
  Arms: 2

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of Xyrem® compared to placebo for the treatment of fibromyalgia in a randomized, double blind, placebo controlled, parallel group trial.

DETAILED DESCRIPTION:
The trial is a randomized, double blind, placebo controlled, parallel group trial in subjects diagnosed with fibromyalgia in accordance with the American College of Rheumatology. Total duration is up to twenty-two (22) weeks of trial participation. Subjects will undergo a screening and withdrawal/washout period lasting up to five (5) weeks combined followed by baseline period lasting one (1) week. Total treatment duration will be fourteen (14) weeks followed by a two week safety follow-up post treatment period. During the screening and withdrawal/washout period, no study medication will be given; however rescue medication up to 4 grams per day of acetaminophen (paracetemol) will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years or older who meet the American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia.

Exclusion Criteria:

* Subjects will be excluded if they have a history of rheumatic disease or other disorders that may compromise reliable representation of subjective symptoms.
* Any other condition that will cause a risk to subjects if they participate in the trial is also a reason for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (116):
- United States (71):
  - East Alabama Arthritis Center, Auburn, Alabama
  - Capstone Clinical Trials, Inc., Birmingham, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - dba 21st Century Neurology, Phoenix, Arizona
  - Orange County Clinical Trials, Anaheim, California
  - Providence Clinical Research, Burbank, California
  - Med Investigations, Inc., Fair Oaks, California
  - North Orange County Research Institute, Inc., Fullerton, California
  - Nerve Pro Research, Irvine, California
  - Northridge Neurological Center, Northridge, California
  - Arroyo Medical Group, Pismo Beach, California
  - Northern California Research, Sacramento, California
  - Sacramento Research Medical Group, Sacramento, California
  - University of CT, Health Center, Farmington, Connecticut
  - Center for Musculoskeletal Pain Research, Gainesville, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Suncoast Internal Medicine Consultants, Largo, Florida
  - AppleMed Research, Miami, Florida
  - Compass Research, Orlando, Florida
  - Clinical Research Group of St. Petersburg, Inc., St. Petersburg, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Lake Rheumatology, Tavares, Florida
  - Center for Arthritis and Rheumatism, Vero Beach, Florida
  - Florida Medical Clinic, P.A., Clinical Research Division, Zephyrhills, Florida
  - Drug Studies America, Marietta, Georgia
  - Coeur d'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Fibromyalgia Treatment Centers of America, Chicago, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Cotton-O'neil Clinical Research center, Topeka, Kansas
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Central Kentucky Research Associates,Inc., Lexington, Kentucky
  - Bluegrass Internal Medicine, Owensboro, Kentucky
  - Louisiana Sleep Foundation, Baton Rouge, Louisiana
  - Capital Clinical Research Associates, Rockville, Maryland
  - Professional Clinical Research at Cyrstal Lake Health Center, Benzonia, Michigan
  - Quest Research Institute, Bingham Farms, Michigan
  - Professional Clinical Research, Cadillac, Michigan
  - Professional Clinical Research at Crystal Lake Health Center, Interlochen, Michigan
  - Arthritis Associates, Hattiesburg, Mississippi
  - Medex Healthcare Research, Inc, St Louis, Missouri
  - St. John's Mercy Health System, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Alan Lichtbroun, MD, East Brunswick, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - North Shore University Hospital, North Shore Pain Services, Valley Stream, New York
  - Great Lakes Medical Research, Westfield, New York
  - Appalachian Regional Medical Associates, Boone, North Carolina
  - Dept of Internal Medicine/Rheumatology The Brody Sch of Medicine at ECU, Greenville, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Health Research Associates, LLC (HRA), Cleveland, Ohio
  - Ohio State U, Immunology/Rheumatology William Davis Medical Research Center, Columbus, Ohio
  - Cleveland Neuro-Sleep Research Institute Inc., Middleburg Heights, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Health Sciences University School of Medicine, Portland, Oregon
  - Tri State Medical Group, Inc., Beaver, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Founders Research, Yardley, Pennsylvania
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Neurology Future Research Trials, Austin, Texas
  - DFW Wellness, Fort Worth, Texas
  - The Methodist Hospital System, Houston, Texas
  - Houston Sleep Center, Houston, Texas
  - R/D Clinical Research, Inc., Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
  - Clinical Health Research, LLC, Sugarland, Texas
  - Arthritis and Osteoporosis Clinic, Research Center of Central Texas, Waco, Texas
  - Alben Goldstein, MD, FACP, Arlington, Virginia
- France (7):
  - Rhumatologie, Amiens
  - CHU de Grenoble-hopital Sud, Échirolles
  - Hopital Claude Huriez Service de medecine Interne, Lille
  - Centre Catherine de Sienne unite d evaluation et de traitment de la douleur CHU Nord, Nantes
  - Hopital Pasteue - Pavillon O, Nice
  - Hopital Hotel Dieu service de medecine interne, Paris
  - CHU Hopital de Rangueil, Toulouse
- Germany (9):
  - Schlosspark-Klinik, Berlin
  - Gemeinschaftspraxis fur Anasthesie und spezielle Schmerztherapie, Böblingen
  - Intensivmedizin der Uniklinik Koln, Cologne
  - Praxis Dr. Wiedeking, Essen
  - Praxis fur Innere Medizin und Rheumatologie, Gräfelfing
  - Gemeinschaftspraxis Schmerzzentrum, Hamburg
  - Rheumazentrum am Krankenhaus Bad Doberan, Hohenfelde - Bad Doberan
  - Praxisklinik Dr. Weiss, Mannheim
  - Praxis Dr. Sohn, Schwalmtal
- Italy (2):
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Pisana-Ospedale Santa Chiara, Pisa
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Mediscch Sprectrum Twente T a.v. Anita mooij-van Dis, Enschede
- Poland (6):
  - Wojewodzki Szpital Zespolony, Elblag
  - Katedra i Klinka Chorob Wewnetrznych i Reumatologii Ortopedyczno-rehabilitacyjny Szpital Kliniczny, Katowice
  - Medycznej w Poznaniu SPZOZ Samodzielny Publiczny Szpital Kliniczny, Poznan
  - w Szczecinie, Szczecinie
  - NZOZ Nasz Lekarz, Torun
  - Instytut Reumatologii, Warsaw
- Spain (9):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Instituto Ferran de Reumatologia, Barcelona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Civil de malaga, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- United Kingdom (10):
  - Barnsley District General Hospital, Rheumatology Department, Barnsley
  - Royal National Hospital for Rheumatic Diseases NHS, Bath
  - Lever Chambers Centre for Health, Bolton
  - King's College London, London
  - 4 West Kennedy Clinical Trial unit, London
  - King College London, London
  - Freeman Hospital, Newcastle
  - Freeman Hospital, Newcastle upon Tyne
  - Philip Arnold Unit, Poole
  - Poole General Hospital, Poole

REFERENCES:
- [Result] Bennett RM, Benson B, Choy EH, Hackshaw KV, Alvarez-Horine S, Wang, YG, Spaeth M. Effects of Sodium Oxybate on Pain, Function, and PGIC in Fibromyalgia: Results From an International, 14-Week, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial. [AAPM abstract 186]. Pain Med. 2010;11(2):317.
- [Result] Swick TJ, Spaeth M, Choy EH, Alvarez-Horine S, Wang YG, Benson B, Bennett R. Sodium Oxybate Reduces Pain and Improves Function and PGIC in Fibromyalgia: Results From an International, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial [AAN abstract P03.293]. Neurology. 2010;74(suppl 2):A280.
- [Result] Bennett RM, Rosenthal N, Lai C, Benson B, Wang YG, Alegre C, Perrot S.. Functionality and Quality of Life Are Improved in Fibromyalgia Patients Treated With Sodium Oxybate: Results From a Phase 3 International Trial. In: American Psychiatric Association New Research Abstracts to the 2010 Annual Meeting; May 22-26, 2010; New Orleans, LA. Abstract NR7-49.
- [Result] Swick TJ, Curtis C, Benson B, Lai C, Wang YG, Rothman J, Sarzi-Puttini P. Fibromyalgia Patients Have Impaired Sleep and Daytime Functioning at Baseline: Data From an International Phase 3 Trial of Sodium Oxybate [APSS abstract 0882]. Sleep. 2010;33(suppl):A295.
- [Result] Swick TJ, Lai C, Benson B, Wang YG, Sarzi-Puttini P. Fibromyalgia Pain, Fatigue, and Sleep Improve With Sodium Oxybate Treatment: A 14-Week Randomized, Double-Blind, Placebo-Controlled International Trial [APSS abstract 0883]. Sleep. 2010;33(suppl):A295.
- [Result] Choy E, Alegre C, Sarzi-Puttini P, van Seventer R, Wang YG, Guinta D, Lai C, Bennett R and the Oxybate in Fibromyalgia 06-009 Study Group. The Effects of Sodium Oxybate on Sleep Disturbance, Fatigue, and Functioning in Fibromyalgia: Results From a Phase 3, Randomized, Double-Blind, Placebo-Controlled International Trial [FRI10411]. Ann Rheum Dis. 2010;69(suppl 3):449.
- [Result] Spaeth M, Perrot S, Samborski W, Bazzichi L, van de Laar M, Guinta D, Wang YG, Lai C, Bennett R and Sodium Oxybate in Fibromyalgia 06-009 Study Group. Sodium Oxybate Treatment Improves Pain, Function, and Patient Global Impression of Change (PGIC) in Fibromyalgia Patients: Results From an International, Randomized, Double-Blind, Placebo-Controlled Trial. Ann Rheum Dis. 2010;69(suppl 3):449

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo taken as two equally divided nightly doses
- Xyrem (Sodium Oxybate) 4.5g: Xyrem 4.5g taken as 2 equally divided nightly doses
- Xyrem (Sodium Oxybate) 6.0g: Xyrem 6.0g taken as 2 equally divided nightly doses
Period: Overall Study
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Started | 188 | 195 | 190
Treated | 188 | 194 | 189
Completed | 131 | 129 | 116
Not Completed | 57 | 66 | 74
Not completed — Adverse Event | 11 | 30 | 40
Not completed — Withdrawal by Subject | 6 | 8 | 5
Not completed — Lost to Follow-up | 5 | 4 | 4
Not completed — Lack of Efficacy | 23 | 18 | 19
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Protocol Violation | 9 | 4 | 4
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Subject started night shift work | 1 | 0 | 0
Not completed — Will start exclusionary medications | 0 | 1 | 0
Not completed — Undergoing tests for Cushings Syndrome | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g | Total
Number analyzed (Participants) | 188 | 195 | 190 | 573
Age Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.73) | 46.6 (10.76) | 46.4 (11.62) | 46.6 (10.72)
Age, Customized [Number; unit: participants]
  18 - 39 years | 43 | 45 | 53 | 141
  40 - 49 years | 62 | 72 | 58 | 192
  50 - 64 years | 81 | 71 | 69 | 221
  >= 65 years | 2 | 7 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 175 | 170 | 513
  Male | 20 | 20 | 20 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 11 | 18 | 39
  White | 173 | 182 | 169 | 524
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 9 | 8 | 7 | 24
  United States | 124 | 123 | 133 | 380
  Poland | 8 | 8 | 6 | 22
  Spain | 18 | 20 | 14 | 52
  Netherlands | 1 | 0 | 3 | 4
  Germany | 22 | 28 | 20 | 70
  Italy | 2 | 4 | 4 | 10
  United Kingdom | 4 | 4 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain VAS (Visual Analog Scale) Response. Percentage of Subjects With a Greater Than or Equal to 30% Reduction in Pain VAS From Baseline (BOCF).
Description: Percentage of pain VAS responders. Subjects with a >= 30% reduction in pain VAS from baseline to endpoint (week 14) were considered responders; all other subjects were considered non-responders. Missing data were handled using BOCF (Baseline Observation Carried Forward). The pain VAS ranges from 0 (no pain) to 100 (worst imaginable pain). The pain VAS was collected morning, afternoon and evening. Baseline is the average value recorded for the measure during the week prior to the end-of-baseline visit. Endpoint is the average value recorded for the measure during the week prior to week 14.
Time Frame: Baseline to Week 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Number analyzed (Participants) | 188 | 195 | 190
Percentage of Participants
  Responder | 20.2 | 35.4 | 35.3
  Non - Responder | 79.8 | 64.6 | 64.7
Statistical Analysis 1: Comparison: Placebo vs Xyrem (Sodium Oxybate) 4.5g vs Xyrem (Sodium Oxybate) 6.0g; Overall Comparison; Test type: Superiority or Other; p = 0.001, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Xyrem (Sodium Oxybate) 4.5g; Pairwise comparison of Xyrem 4.5g and placebo; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Xyrem (Sodium Oxybate) 6.0g; Pairwise comparison of Xyrem 6.0g and placebo; Test type: Superiority or Other; p = 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Serious Adverse Events (participants affected / at risk) | 3/188 | 2/194 | 3/189
Other Adverse Events (participants affected / at risk) | 126/188 | 146/194 | 156/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=188) | Xyrem (Sodium Oxybate) 4.5g (N=194) | Xyrem (Sodium Oxybate) 6.0g (N=189)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Secondary Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=188) | Xyrem (Sodium Oxybate) 4.5g (N=194) | Xyrem (Sodium Oxybate) 6.0g (N=189)
Palpatations (Cardiac disorders) | 2 | 2 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 8 | 7
Vision Blurred (Eye disorders) | 2 | 4 | 3
Nausea (Gastrointestinal disorders) | 16 | 37 | 40
Diarrhoea (Gastrointestinal disorders) | 15 | 14 | 22
Vomiting (Gastrointestinal disorders) | 6 | 10 | 16
Constipation (Gastrointestinal disorders) | 3 | 5 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2 | 5
Dry Mouth (Gastrointestinal disorders) | 2 | 2 | 6
Abdominal Pain (Gastrointestinal disorders) | 2 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 4
Fatigue (General disorders) | 4 | 6 | 11
Oedema Peripheral (General disorders) | 4 | 3 | 12
Pain (General disorders) | 2 | 4 | 2
Malaise (General disorders) | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 7 | 13 | 13
Influenza (Infections and infestations) | 12 | 4 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 6 | 4
Sinusitis (Infections and infestations) | 5 | 5 | 1
Weight Increased (Investigations) | 1 | 4 | 3
Blood Pressure Increased (Investigations) | 0 | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 1 | 7 | 4
Decrease Appetite (Metabolism and nutrition disorders) | 0 | 2 | 4
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 | 7 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 8 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 9
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Headache (Nervous system disorders) | 36 | 41 | 43
Dizziness (Nervous system disorders) | 3 | 23 | 25
Somnolence (Nervous system disorders) | 3 | 7 | 11
Paraesthesia (Nervous system disorders) | 5 | 4 | 9
Migraine (Nervous system disorders) | 6 | 3 | 2
Tremor (Nervous system disorders) | 0 | 6 | 3
Disturbance in Attention (Nervous system disorders) | 1 | 4 | 2
Insomnia (Psychiatric disorders) | 6 | 15 | 8
Anxiety (Psychiatric disorders) | 3 | 10 | 15
Depression (Psychiatric disorders) | 0 | 3 | 5
Disorientation (Psychiatric disorders) | 1 | 2 | 5
Confusional State (Psychiatric disorders) | 0 | 1 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Hypertension (Vascular disorders) | 3 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other